CLINICAL TRIAL: NCT06978803
Title: HYEEG Discourse in Psychosis: A Neurobehavioural Study
Acronym: DISCOURSE-NB
Status: Recruiting | Type: Observational
Sponsor: Douglas Mental Health University Institute (Other)
Responsible Party: Principal Investigator, Lena Palaniyappan, Professor of Psychiatry, Douglas Mental Health University Institute
Other Study IDs: 2023-595
Record Dates: First submitted 2025-01-13; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-11

CONDITIONS: Psychosis; Schizophrenia Disorders
Keywords: hyperscanning eeg; psychosis; imitation tasks; interbrain synchrony; motor imitation; motor behaviour; speech disorganization; natural language processing
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy controls: 1. English or French-speaking participants (as dyads matched for language preference).
  2. Ages 18-60 years.
  3. No diagnosis of schizophrenia or schizoaffective illness based on the Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 criteria.
- Patients: 1. English or French-speaking participants (as dyads matched for language preference).
  2. Ages 18-60 years.
  3. Patients meeting the operational criteria for schizophrenia or schizoaffective illness as previously diagnosed by their treating psychiatrist, based on the Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 criteria.
  4. Patients with less than 5 years of illness onset, based on the time of starting treatment with antipsychotic medication.

SUMMARY:
This multimodal study explores the mechanisms underlying social dysfunction in individuals with schizophrenia. It focuses on the relationship between disorganized communication and social interaction, aiming to identify measurable markers of disorganized communication and link them to clinical symptoms and social functioning.

Key Research Questions:

How do neural and behavioural synchrony contribute to social impairments in schizophrenia?

What roles do interbrain synchrony, motor imitation, reaction time, and verbal coherence play in disorganized communication?

Participants will:

1. Engage in structured and semi-structured real-time social interactions while undergoing dual-brain electroencephalogram (EEG) hyperscanning to measure neural and behavioural activity.
2. Perform nonverbal tasks such as motor imitation and reaction time assessments to investigate coordination and behavioural synchrony patterns.
3. Participate in a clinical interview that evaluates verbal production, thought coherence, and speech organization.

By combining these assessments, the study aims to advance our understanding of how social and communication impairments manifest in schizophrenia. The findings will contribute to developing improved diagnostic tools and targeted interventions, ultimately supporting patients in achieving better social functioning and quality of life.

DETAILED DESCRIPTION:
INTRODUCTION

Schizophrenia, often associated with psychosis, is a severe mental disorder that profoundly impacts individuals, families, and society, diminishing quality of life and well-being globally. Disorganized communication-a hallmark feature of schizophrenia-is characterized by impairments in speech production, gesture-speech coordination, and motor behaviours that disrupt the ability to convey and interpret meaning in social contexts. These deficits profoundly undermine interpersonal relationships and social connectedness, creating barriers to meaningful social engagement. The impact of these challenges is particularly acute among marginalized populations, who face additional systemic obstacles such as stigma, reduced access to healthcare, and limited social support networks.

The early onset of psychosis, typically during late adolescence or early adulthood, coincides with a critical developmental period marked by heightened neuroplasticity. Social preferences, communication patterns, and adaptive behaviours are formed during this period. This developmental window is particularly vulnerable to disruptions in social interactions, which can derail neurobehavioural trajectories and contribute to long-term social dysfunction. Understanding how disorganized communication emerges and persists during this critical window is essential for designing early interventions to mitigate its effects.

Social disconnection-the breakdown of interpersonal connectivity and adaptability-is likely rooted in disruptions to the underlying neurobehavioural dynamics that facilitate coordinated interpersonal interactions. These dynamics include synchrony in speech, movement, and neural activity, which are crucial for effective social functioning. Despite significant advancements in mental health research, the specific neural and behavioural underpinnings of disorganized communication remain poorly understood, particularly in their relationship to broader social dysfunction in schizophrenia.

Addressing these challenges requires advanced tools capable of capturing the dynamic and reciprocal processes underlying social interactions. Real-time electroencephalogram (EEG) hyperscanning offers a robust method for studying interbrain synchrony, a critical interpersonal dynamic essential for coordinated social behaviour. This technique allows for the simultaneous recording of brain activity from two individuals engaged in reciprocal sensorimotor interactions, such as cooperative imitation. By analyzing patterns of synchrony and desynchrony in interbrain activity and associated bodily dynamics, EEG hyperscanning provides a detailed framework for examining the mechanisms underlying nonverbal communication and its disruptions.

This study integrates a speech elicitation protocol with standardized transcription methods and natural language processing (NLP) techniques developed by the Diverse International Scientific Consortium for Research in Thought, Language and Communication in Psychosis group. Additionally, it incorporates a validated motor imitation protocol from prior research with healthy participants. By combining EEG hyperscanning data with detailed analyses of verbal and nonverbal behaviours, the study seeks to identify disruptions in cooperative imitation and their links to speech disorganization, providing new insights into the mechanisms of disorganized communication.

This research aims to elucidate the mechanisms underlying disorganized communication by linking neural synchrony to verbal coherence, motor synchrony, and other neurobehavioural responses. These findings aim to inform the development of targeted early interventions that address both the behavioural and neural dimensions of disorganized communication in individuals with psychosis.

RATIONALE

The frontal and temporoparietal brain regions play critical roles in selective attention, inhibitory control, and social cognition. In schizophrenia, disruptions in neural synchronization between these regions-particularly within the alpha (8-12 Hz), beta (13-30 Hz), and gamma (30-100 Hz) frequency bands-are well-documented. Impaired functional connectivity between the prefrontal cortex and temporoparietal regions may contribute to maladaptive, self-focused attention, impairing the processing and integration of external social cues.

Specific dysregulations are hypothesized to underlie these deficits: alpha-band disruptions weaken attentional filtering, beta-band abnormalities impair sustained cognitive control, and gamma-band deficits disrupt the integration of social and perceptual information. These disruptions are expected to create an imbalance between internal and external processing, reducing neural coherence and phase synchronization during social exchanges. This breakdown in neural and behavioural coordination is hypothesized to manifest as neurobehavioural markers of disorganized communication-a hallmark feature of schizophrenia.

SPECIFIC HYPOTHESES

1. Impairments in Inhibition-Based Imitation:

   Patients with schizophrenia will exhibit significant impairments in inhibition-based imitation compared to automatic imitation, as the former requires higher cognitive control. These impairments are expected to reflect deficits in executive function, particularly the ability to selectively suppress automatic responses.
2. Correlation Between Imitation and Speech Disorganization:

   Difficulties in inhibition-based imitation will positively correlate with the severity of speech disorganization. Speech disorganization will be measured through clinical evaluations, structured interviews, and natural language processing (NLP) analyses, highlighting shared neural mechanisms underlying executive function and social communication.
3. Reduced Interbrain Synchrony:

Interbrain synchrony during interpersonal coordination, assessed using EEG hyperscanning and behavioural analysis, will be significantly reduced in patients compared to healthy controls. This reduction is expected to reflect disruptions in neural oscillations critical for effective social interaction.

MULTIMODAL ANALYSES AND FUTURE DIRECTIONS

This research employs multimodal exploratory analyses to investigate the relationships between interbrain synchrony, bodily activity measures, and conversational speech variables, such as verbal coherence and semantic similarity. These analyses will also explore how these measures relate to symptom severity, providing a comprehensive understanding of their interplay.

By quantifying the effect sizes of these relationships, the study aims to establish foundational evidence for the development of larger-scale research. The results are expected to inform the refinement of experimental protocols, identify robust biomarkers of social dysfunction, and guide the design of targeted early interventions for individuals with psychosis.

ELIGIBILITY:
Inclusion Criteria:

1. English or French-speaking participants (as dyads matched for language preference).
2. Ages 18-60 years.
3. Patients meeting the operational criteria for schizophrenia or schizoaffective illness as previously diagnosed by their treating psychiatrist, based on the Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 criteria (Zipursky et al., 2020).
4. Patients with less than 5 years of illness onset, based on the time of starting treatment with antipsychotic medication.

Exclusion Criteria:

1. Participants should not have a primary diagnosis of Alcohol or Drug abuse or addiction (however, co-morbid substance abuse with a primary diagnosis of psychotic disorder is not an exclusion criterion).
2. Participants should not have a severe medical disorder that would explain psychotic symptoms.
3. Participants should not have a past or current history of a primary neurological disorder that can affect speech output
4. Participants with IQ below 70 or a concurrent pervasive developmental disorder (e.g., autism) will also be excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with psychosis will be recruited from the following Douglas Mental Health University Institute areas: l'Étape Outpatient Clinic, Assertive Community Treatment Clinics, Intensive Psychosocial Rehab Clinic, and the Prevention and Early Intervention Program for Psychosis (PEPP) clinics in CIUSSS de l'ouest-de-L'île-de-Montréal, in association with the Centre for Youth Mental Health at the Douglas. Healthy Control participants will be recruited from the Greater Montreal Area using online study advertisements (Facebook, Kijiji, Twitter) and research study posters placed on bulletin boards.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-10-22 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Inter-brain phase synchronization using Phase Locking Index via hyperscanning during communication | baseline
  Using oscillatory and time-frequency analyses of electroencephalography (EEG) hyperscanning data, inter-brain synchronization will be calculated via phase locking value for both patients and control subjects. This value will be related to: (1) verbal data from clinical interviews analyzed using Natural Language Processing techniques, including sentiment analysis to assess emotional tone, coherence classification to evaluate logical flow, and semantic similarity analysis (2) nonverbal measures such as motor synchrony, imitation accuracy, and reaction time.

OTHER OUTCOMES:
Composite Index of Severity as Measured by the Positive and Negative Syndrome Scale (PANSS), THought and Language Index and Social and Occupational Functioning (SOFAS) | baseline
  This composite outcome will be a single factor score; higher values will reflect more severe symptoms and poor social functioning. Lower values will reflect better functioning and less severe symptoms. This will be derived from factor analysis of Positive and Negative Syndrome Scale (PANSS), Social and Occupational Functioning Assessment Scale (SOFAS), and the scores from the Thought and Language Index (TLI) clinical interview. This will be related to the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Lena Palaniyappan, MD, PhD, Principal Investigator — Douglas Mental Health University Institute
Locations (1):
- Douglas Mental Health University Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
We propose to use a clinical linguistic archiving system called the TalkBank (https://www.talkbank.org/) for data sharing purposes. TalkBank registry/database is located at Carnegie Mellon University, Pittsburgh, Pennsylvania-USA. Several filters are used to de-identify the recorded speech data before storage in the databank. Firstly, the Discourse protocol explicitly avoids using proper nouns and names/addresses. Second, the transcribed data is checked, and any proper names are replaced by common names (e.g., 'McGill' will be changed to 'University') or bleeped out (for audio data). If requested, we will play back the recorded responses to check if the participant is comfortable with the degree of anonymity. Identifying demodemographics will not be stored alongside the speech data to reduce triangulation. Finally, sharing is controlled by password protection, and a re-review is done to remove identifying information before sharing is initiated.
Supporting Information: Study Protocol
Time Frame: December 2028 for an unlimitied amount of time. There are no plans for data destruction of the study information stored (de-identified audio and transcriptions) within TalkBank.
Access Criteria: The anonymized speech data will be retained on an access-controlled secure database hosted by TalkBank. We anticipate this being available within 2 years of the enrolment of the last participant. For more information see https://psychosis.talkbank.org/ and https://discourseinpsychosis.org/

REFERENCES:
- [Background] Rybarczyk, B., Social and Occupational Functioning Assessment Scale (SOFAS), in Encyclopedia of Clinical Neuropsychology, J.S. Kreutzer, J. DeLuca, and B. Caplan, Editors. 2011, Springer New York: New York, NY. p. 2313-2313.
- [Background] Liechti S, Capodilupo G, Opler DJ, Opler M, Yang LH. A Developmental History of the Positive and Negative Syndrome Scale (PANSS). Innov Clin Neurosci. 2017 Dec 1;14(11-12):12-17. PMID 29410932
- [Background] Tang SX, Kriz R, Cho S, Park SJ, Harowitz J, Gur RE, Bhati MT, Wolf DH, Sedoc J, Liberman MY. Natural language processing methods are sensitive to sub-clinical linguistic differences in schizophrenia spectrum disorders. NPJ Schizophr. 2021 May 14;7(1):25. doi: 10.1038/s41537-021-00154-3. PMID 33990615
- [Background] Morgan SE, Diederen K, Vertes PE, Ip SHY, Wang B, Thompson B, Demjaha A, De Micheli A, Oliver D, Liakata M, Fusar-Poli P, Spencer TJ, McGuire P. Natural Language Processing markers in first episode psychosis and people at clinical high-risk. Transl Psychiatry. 2021 Dec 13;11(1):630. doi: 10.1038/s41398-021-01722-y. PMID 34903724
- [Background] Liddle PF, Ngan ET, Caissie SL, Anderson CM, Bates AT, Quested DJ, White R, Weg R. Thought and Language Index: an instrument for assessing thought and language in schizophrenia. Br J Psychiatry. 2002 Oct;181:326-30. doi: 10.1192/bjp.181.4.326. PMID 12356660
- [Background] Kinreich S, Djalovski A, Kraus L, Louzoun Y, Feldman R. Brain-to-Brain Synchrony during Naturalistic Social Interactions. Sci Rep. 2017 Dec 6;7(1):17060. doi: 10.1038/s41598-017-17339-5. PMID 29213107
- [Background] Dumas G, Nadel J, Soussignan R, Martinerie J, Garnero L. Inter-brain synchronization during social interaction. PLoS One. 2010 Aug 17;5(8):e12166. doi: 10.1371/journal.pone.0012166. PMID 20808907
- [Background] Czeszumski A, Eustergerling S, Lang A, Menrath D, Gerstenberger M, Schuberth S, Schreiber F, Rendon ZZ, Konig P. Hyperscanning: A Valid Method to Study Neural Inter-brain Underpinnings of Social Interaction. Front Hum Neurosci. 2020 Feb 28;14:39. doi: 10.3389/fnhum.2020.00039. eCollection 2020. PMID 32180710
- [Background] Carollo A, Esposito G. Hyperscanning literature after two decades of neuroscientific research: A scientometric review. Neuroscience. 2024 Jul 23;551:345-354. doi: 10.1016/j.neuroscience.2024.05.045. Epub 2024 Jun 10. PMID 38866073
- [Background] Hirano Y, Uhlhaas PJ. Current findings and perspectives on aberrant neural oscillations in schizophrenia. Psychiatry Clin Neurosci. 2021 Dec;75(12):358-368. doi: 10.1111/pcn.13300. Epub 2021 Oct 29. PMID 34558155
- [Background] Geng JJ, Vossel S. Re-evaluating the role of TPJ in attentional control: contextual updating? Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 2):2608-20. doi: 10.1016/j.neubiorev.2013.08.010. Epub 2013 Aug 30. PMID 23999082
- [Background] daSilva EB, Wood A. How and Why People Synchronize: An Integrated Perspective. Pers Soc Psychol Rev. 2025 May;29(2):159-187. doi: 10.1177/10888683241252036. Epub 2024 May 21. PMID 38770754
- [Background] Liu T, Pelowski M. Clarifying the interaction types in two-person neuroscience research. Front Hum Neurosci. 2014 Apr 30;8:276. doi: 10.3389/fnhum.2014.00276. eCollection 2014. No abstract available. PMID 24817848
- [Background] Nowak A, Vallacher RR, Zochowski M, Rychwalska A. Functional Synchronization: The Emergence of Coordinated Activity in Human Systems. Front Psychol. 2017 Jun 13;8:945. doi: 10.3389/fpsyg.2017.00945. eCollection 2017. PMID 28659842
- [Background] Koul A, Ahmar D, Iannetti GD, Novembre G. Interpersonal synchronization of spontaneously generated body movements. iScience. 2023 Feb 1;26(3):106104. doi: 10.1016/j.isci.2023.106104. eCollection 2023 Mar 17. PMID 36852275
- [Background] Bolis D, Dumas G, Schilbach L. Interpersonal attunement in social interactions: from collective psychophysiology to inter-personalized psychiatry and beyond. Philos Trans R Soc Lond B Biol Sci. 2023 Feb 13;378(1870):20210365. doi: 10.1098/rstb.2021.0365. Epub 2022 Dec 26. PMID 36571122
- [Background] Schilbach L. Towards a second-person neuropsychiatry. Philos Trans R Soc Lond B Biol Sci. 2016 Jan 19;371(1686):20150081. doi: 10.1098/rstb.2015.0081. PMID 26644599
- [Background] Green MF, Horan WP, Lee J. Nonsocial and social cognition in schizophrenia: current evidence and future directions. World Psychiatry. 2019 Jun;18(2):146-161. doi: 10.1002/wps.20624. PMID 31059632
- [Background] Gil-Berrozpe GJ, Peralta V, Sanchez-Torres AM, Moreno-Izco L, Garcia de Jalon E, Peralta D, Janda L, Cuesta MJ; SEGPEPs group. Psychopathological networks in psychosis: Changes over time and clinical relevance. A long-term cohort study of first-episode psychosis. Schizophr Res. 2023 Feb;252:23-32. doi: 10.1016/j.schres.2022.12.046. Epub 2023 Jan 6. PMID 36621323
- [Background] Rotenberg M, Tuck A, Anderson KK, McKenzie K. The Incidence of Psychotic Disorders and Area-level Marginalization in Ontario, Canada: A Population-based Retrospective Cohort Study. Can J Psychiatry. 2022 Mar;67(3):216-225. doi: 10.1177/07067437211011852. Epub 2021 Apr 26. PMID 33896210
- [Background] Jongsma HE, Turner C, Kirkbride JB, Jones PB. International incidence of psychotic disorders, 2002-17: a systematic review and meta-analysis. Lancet Public Health. 2019 May;4(5):e229-e244. doi: 10.1016/S2468-2667(19)30056-8. PMID 31054641
- [Background] Green MF, Horan WP, Lee J, McCleery A, Reddy LF, Wynn JK. Social Disconnection in Schizophrenia and the General Community. Schizophr Bull. 2018 Feb 15;44(2):242-249. doi: 10.1093/schbul/sbx082. PMID 28637195
- [Background] Correll CU, Solmi M, Croatto G, Schneider LK, Rohani-Montez SC, Fairley L, Smith N, Bitter I, Gorwood P, Taipale H, Tiihonen J. Mortality in people with schizophrenia: a systematic review and meta-analysis of relative risk and aggravating or attenuating factors. World Psychiatry. 2022 Jun;21(2):248-271. doi: 10.1002/wps.20994. PMID 35524619
- [Background] Olarewaju E, Dumas G, Palaniyappan L. Disorganized Communication and Social Dysfunction in Schizophrenia: Emerging Concepts and Methods. Curr Psychiatry Rep. 2023 Nov;25(11):671-681. doi: 10.1007/s11920-023-01462-4. Epub 2023 Sep 23. PMID 37740852
- [Background] Cotter J, Granger K, Backx R, Hobbs M, Looi CY, Barnett JH. Social cognitive dysfunction as a clinical marker: A systematic review of meta-analyses across 30 clinical conditions. Neurosci Biobehav Rev. 2018 Jan;84:92-99. doi: 10.1016/j.neubiorev.2017.11.014. Epub 2017 Nov 24. PMID 29175518
- [Background] Gur RC, Gur RE. Social cognition as an RDoC domain. Am J Med Genet B Neuropsychiatr Genet. 2016 Jan;171B(1):132-41. doi: 10.1002/ajmg.b.32394. Epub 2015 Nov 26. PMID 26607670
- [Background] Porcelli S, Van Der Wee N, van der Werff S, Aghajani M, Glennon JC, van Heukelum S, Mogavero F, Lobo A, Olivera FJ, Lobo E, Posadas M, Dukart J, Kozak R, Arce E, Ikram A, Vorstman J, Bilderbeck A, Saris I, Kas MJ, Serretti A. Social brain, social dysfunction and social withdrawal. Neurosci Biobehav Rev. 2019 Feb;97:10-33. doi: 10.1016/j.neubiorev.2018.09.012. Epub 2018 Sep 20. PMID 30244163
- [Background] Kennedy DP, Adolphs R. The social brain in psychiatric and neurological disorders. Trends Cogn Sci. 2012 Nov;16(11):559-72. doi: 10.1016/j.tics.2012.09.006. Epub 2012 Oct 6. PMID 23047070
- See also: Related Info — https://ceymh-cesmj.ca/research/
- See also: Related Info — https://douglas.research.mcgill.ca/clinical_studies/discourse-in-psychosis-a-neurobehavioural-study/